CLINICAL TRIAL: NCT06859957
Title: Melatonin for Patients With Chronic Low Back Pain - a Randomized Placebo-controlled Trial
Brief Title: Melatonin for Patients With Chronic Low Back Pain
Acronym: MELBACK
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bart Koes (Other)
Responsible Party: Sponsor-Investigator, Bart Koes, Prof. dr., Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PaNaMa 11825; 2024-514769-20-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-31; First posted 2025-03-05 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-03

CONDITIONS: Chronic Low-back Pain (cLBP)
Keywords: Chronic low back pain; Melatonin
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Melatonin (Experimental): 10mg of melatonin daily for a period of 6 weeks
  Interventions: Drug: Melatonin 10 mg

INTERVENTIONS:
Drug: Melatonin 10 mg — 10 mg melatonin daily for a period of 6 weeks
  Arms: Melatonin
Drug: Placebo — Daily placebo for a period of 6 weeks
  Arms: Placebo

SUMMARY:
Low back pain is one of the conditions causing more disability worldwide. The use of pain medications is substantial in patients with chronic LBP. But the efficacy of commonly used analgesics is modest. More than half of patients with chronic LBP also has sleep problems. In recent years, some preliminary studies have shown a promising effect of melatonin for the treatment of pain.

The objective of this study is to investigate the efficacy of melatonin, relative to placebo, in patients with chronic LBP.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65
* understand and write Dutch
* LBP for 3 months or longer
* LBP must be present on 'most days' or 'every day' within the past 3 months
* LBP must limit life or work activities on 'some days', 'most days', or 'every day' within the past 3 months
* average LBP intensity of ≥4 on a 0-10 NRS in the past 7 days

Exclusion Criteria:

* LBP resulting from a specific cause such as malignancy, fracture, lumbar radiculopathy and spinal stenosis
* Radiating pain into the leg that goes further (down) than the knee
* Inflammatory/autoimmune arthritis
* Severe physical or psychiatric co-morbidities
* Contraindications to melatonin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in low back pain intensity | from baseline to end of treatment at 6 weeks
  Change in low back pain intensity (average pain intensity past 7 days), measured on a 0-10 Numeric Rating Scale (NRS) where 0 means no pain and 10 means worst pain imaginable, from baseline to 6 weeks

SECONDARY OUTCOMES:
Back pain-related disability (RMDQ) | baseline to end of treatment at 6 weeks and 3 months and 6 months follow-up
  Back pain-related disability is measured using the Roland Morris Disability Questionnaire (RMDQ). The RMDQ outcome ranges from 0-24, where a higher score means more disability.
Global perceived effect score | baseline to end of treatment at 6 weeks and 3 months and 6 months follow-up
  Using Global perceived effect (GPE) questionnaire (7-point scale), where a score of 1 means highly satisfied/ great recovery and a score of 7 means highly dissatisfied / poor recovery.
Physical and mental health measured using the PROMIS Global Health | baseline to end of treatment at 6 weeks and 3 months and 6 months follow-up
  Physical and mental health measured using the PROMIS Global Health questionnaire.
  A 10 items questionnaire, items are scored from 1-5 where a score of 5 is the best outcome and a score of 1 is the worst outcome.
Health related quality of life measured using the EQ-5D-5L | baseline to end of treatment at 6 weeks and 3 months and 6 months follow-up
  Measured using the EQ-5D-5L (questionnaire).
  The EQ-5D-5L consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS (0-100) records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
Insomnia measured using the Insomnia Severity Index | baseline to end of treatment at 6 weeks and 3 months and 6 months follow-up
  Measured using the Insomnia Severity Index (ISI) (questionnaire). The questionnaire consists of 7 questions, all scored with a score ranging from 0-3. The total score ranges from 0 (no sleeping problems) to 28 (severe sleeping problems)
Self-reported number of days with sick leave | baseline to 3 months and 6 months follow-up
  Using a questionnaire
Emotional functioning using the Beck Depression Inventory (BDI) | baseline to end of treatment at 6 weeks
  Measured using the Beck Depression Inventory (BDI) (questionnaire). A 21-item questionnaire, every item is scored from 0-3. This leads to a total score from 0 (best outcome) to 63 (worst outcome)
Pain-related anxiety measured using the Pain Anxiety Symptoms Scale | baseline to end of treatment at 6 weeks
  Measured using the Pain Anxiety Symptoms Scale (PASS) (questionnaire). A 40-item questionnaire (ranging from 0-200), where a high score means high pain related anxiety.
Neuropathic pain measured using PainDETECT | baseline to end of treatment at 6 weeks and 3 months and 6 months follow-up
  Measured using PainDETECT (questionnaire). A 9-item questionnaire, with 7 weighted descriptor items (from never to very strongly) and 2 items related to spatial and temporal pain characteristics.
  A total score of 19 or more is indicative of likely neuropathic pain.
Productivity losses measured using iMTA Productivity Cost Questionnaire | baseline to 3 months and 6 months follow-up
  iMTA Productivity Cost Questionnaire is used. The questionnaire consists of 18 questions in total. To calculate the costs of production losses, volumes are multiplied by unit costs.
Direct costs of medical care measured using iMCQ Medical Consumption Questionnaire | baseline to 3 months and 6 months follow-up
  Direct costs of medical care measured using iMCQ Medical Consumption Questionnaire.
  The questionnaire consists of 29 items. Questions are answered with yes/no, or participants are asked to fill in a number, for example "How many appointments with the physiotherapist did you have in the past 3 months?". The costs of medical consumption are calculated by multiplying measured volumes of care by the cost price per unit of care.
Adverse events | baseline to end of treatment at 6 weeks and 3 months and 6 months follow-up
  Using questionnaire according to the Common Terminology Criteria for Adverse Events (CTCAE)

OTHER OUTCOMES:
Activity patterns measured using a GENEActiv activity tracker | 7 days during treatment period
  A GENEActiv activity tracker is worn for a period of 7 days during the 6-week treatment period by a subgroup of 60 participants. This device can measure activity and sleep. This measure is use as an explorative objective and only descriptive statistics of the data will be given. GENEActiv software is used to analyse the data.
Sleep reports measured using a GENEActiv activity tracker | 7 days during treatment period
  A GENEActiv activity tracker is worn for a period of 7 days during the 6-week treatment period by a subgroup of 60 participants. This device can measure activity and sleep. A sleep report is created using the GENEActiv software. This measure is used as an explorative measure, only descriptive statistics are done.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, Netherlands